CLINICAL TRIAL: NCT06333717
Title: Impact of Whole Grain Rye Bread on Modulating Microbiota-gut-brain Axis in Healthy Subjects
Brief Title: Impact of Whole Grain Rye Bread on Health
Acronym: FBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Örebro University, Sweden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Dnr 2020-03709
Record Dates: First submitted 2024-02-28; First posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Healthy Diet
Keywords: dietary fibre; microbiota; gut-brain axis

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double blinding
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-fibre bread (Experimental): Six slices (180 g) of whole grain rye bread divided over the meals during the day for 3 weeks
  Interventions: Dietary Supplement: Whole grain bread
- Control bread (Placebo Comparator): Six slices (180 g) of control bread containing refined wheat and oat flour divided over the meals during the day for 3 weeks
  Interventions: Dietary Supplement: Control bread

INTERVENTIONS:
Dietary Supplement: Whole grain bread — Consumption of high-fibre bread as a dietary supplementation
  Arms: High-fibre bread
Dietary Supplement: Control bread — Consumption of control bread as a dietary supplementation
  Arms: Control bread

SUMMARY:
This randomized controlled trial aims to study how a high intake of a fibre-rich bread affects the composition and functioning of the gut microbiota in healthy subjects, and how this, in turn, impacts on the release of gut peptides, intestinal permeability, stress and cognitive performance.

DETAILED DESCRIPTION:
Healthy subjects will be recruited for a 3-week, randomized, parallel-controlled study. Subjects that are eligible to take part in the study will be blinded and randomly allocated to consume a fibre-rich bread or a control bread daily for 3 weeks. Measurements of biomarkers related to the gut-brain axis, microbiota composition and functioning, intestinal permeability, stress and cognitive functioning will be conducted on two separate test days, at baseline and after the 3 weeks intervention. On both test days (day 0 and day 21) subjects will come to the study centre after a 10 hours overnight fast and will deliver faecal samples collected at home. At the study centre, blood samples will be collected and a device for continuous assessment of autonomic nervous system response (Biopac) will be placed. Subjects will drink a multisugar solution and urine samples will be collected for gut permeability analysis. Sugar solution intake will be followed by a baseline period during which participants will rest for 30 minutes to adapt to the laboratory setting. After the baseline period, subjects will conduct a stress test and cognitive tests. Visual analogue scales (VAS) to assess momentary perceived stress levels and saliva samples will be collected before and after the stress test. The study subjects will also complete questionnaires at both visits (food frequency questionnaire, food diary, physical activity, gastrointestinal symptom rating scale, Euro Quality of Life).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-44 years
* Body mass index (BMI) 18,5-30 kg/m2 (normal weight or overweight)

Exclusion Criteria:

* Significant acute or chronic illness, including an inflammatory or a functional disease of gastrointestinal track and psychiatric and psychological disorders
* Anxiety or depression (according to Hospital Anxiety and Depression Scale (HADS score) and Depression Anxiety Stress Scale (DASS-21 score))
* Use of a medication that may interfere with the study (e.g. cannabis, antipsychotics, anxiolytics, antidepressants, proton-pump inhibitors)
* Abuse of alcohol or drugs (according to AUDIT score)
* Use of antibiotic medication within the past 3 months before the study
* Use of laxative or anti-diarrhoea medication within the past 3 months before the study
* Regular consumption of probiotic or prebiotic product for the past 6 weeks before the study
* A diet that may interfere with the study (such as gluten free or low-carb diet)
* Smoking
* Pregnancy or breastfeeding
* Premenopausal female with irregular or short menstruation cycle and not using hormonal contraception
* Colour blindness, dyslexia or dyscalculia
* Unable to absent from caffeine, alcohol or intense exercise for 12 hours prior measurements.

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2021-03-03 (Actual); Study Completion 2021-11-05 (Actual)

PRIMARY OUTCOMES:
Microbiota composition baseline vs after intervention using 16S RNA gene sequencing | faecal samples collected before and after intake of bread for 3 weeks
  Difference in gut microbiota composition in faecal samples before (baseline) and after intake of six slices of bread for 3 weeks (after intervention) using 16S RNA gene sequencing

SECONDARY OUTCOMES:
Microbiota composition whole grain rye bread vs control bread using 16S RNA gene sequencing | faecal samples collected before and after intake of bread for 3 weeks
  Difference in gut microbiota composition in faecal samples between the study arms using 16S RNA gene sequencing
Concentrations of circulatory short-chain fatty acids SCFA | blood samples collected before and after intake of bread for 3 weeks
  Difference in blood levels of SCFA between and within intervention groups after intake of bread for 3 weeks
Concentrations of faecal SCFA | faecal samples collected before and after intake of bread for 3 weeks
  Difference in faecal levels of SCFA between and within intervention groups after intake of bread for 3 weeks
Concentrations of blood glucagon like peptide-1 (GLP-1) | blood samples collected before and after intake of bread for 3 weeks
  Difference in blood levels of GLP-1 between and within intervention groups after intake of bread for 3 weeks
Concentrations of blood glucagon like peptide-2 (GLP-2) | blood samples collected before and after intake of bread for 3 weeks
  Difference in blood levels of GLP-2 between and within intervention groups after intake of bread for 3 weeks
Concentrations of blood peptide YY (PYY) | blood samples collected before and after intake of bread for 3 weeks
  Difference in blood levels of PYY between and within intervention groups after intake of bread for 3 weeks
Concentrations of blood gastric inhibitory polypeptide (GIP) | blood samples collected before and after intake of bread for 3 weeks
  Difference in blood levels of GIP between and within intervention groups after intake of bread for 3 weeks
Concentrations of blood neuroactive peptide Y (NPY) | blood samples collected before and after intake of bread for 3 weeks
  Difference in blood levels of NPY between and within intervention groups after intake of bread for 3 weeks
Concentrations of blood brain-derived neurotrophic factor (BDNF) | blood samples collected before and after intake of bread for 3 weeks
  Difference in blood levels of BDNF between and within intervention groups after intake of bread for 3 weeks
Concentrations of blood cytokines | blood samples collected before and after intake of bread for 3 weeks
  Difference in blood levels of cytokines between and within intervention groups after intake of bread for 3 weeks
Concentrations of blood alkylresorcinols | blood samples collected before and after intake of bread for 3 weeks
  Difference in blood levels of alkylresorcinols between and within intervention groups after intake of bread for 3 weeks
Concentrations of blood lipopolysaccharide-binding protein (LBP) | blood samples collected before and after intake of bread for 3 weeks
  Difference in blood levels of LBP between and within intervention groups after intake of bread for 3 weeks
Concentrations of blood soluble CD-14 (sCD-14) | blood samples collected before and after intake of bread for 3 weeks
  Difference in blood levels of sCD-14 between and within intervention groups after intake of bread for 3 weeks
Concentrations of sugars in urine | urine samples collected before and after intake of bread for 3 weeks
  Difference on intestinal permeability between and within intervention groups after intake of bread for 3 weeks measured by the excretion of sugars contained in a multi-sugar solution
Concentrations of saliva cortisol during stress test | Saliva samples collected before the stress test, after the introduction phase, directly after the acute stress phase, 5 minutes, 10-15 minutes, 60 minutes, and 75 minutes after the stress test
  Difference in saliva levels of cortisol produced during stress test between and within intervention groups after intake of bread for 3 weeks
Concentrations of saliva alpha-amylase during stress test | Saliva samples collected before the stress test, after the introduction phase, directly after the acute stress phase, 5 minutes, 10-15 minutes, 60 minutes, and 75 minutes after the stress test
  Difference in saliva levels of a-amylase produced during stress test between and within intervention groups after intake of bread for 3 weeks

OTHER OUTCOMES:
Gastrointestinal symptoms measured by Gastrointestinal Symptom Rating Scale in Irritable Bowel Syndrome (GSRS-IBS) | 3 weeks
  Difference in the frequency and severity of gastrointestinal symptoms between and within intervention groups after the intake of bread for 3 weeks. The GSRS-IBS contains 13 self-report items rated on a 6-point Likert scale ranging from 1 (no discomfort at all) to 7 (very severe discomfort). Total scores range from 0 to 78.
Food habits measured by an electronic food frequency questionnaire Mealq | 3 weeks
  Survey of participants' food habits before and during the intake of bread for 3 weeks
Food habits measured by a Food diary | 3 days
  Survey of participants' food habits before and during the intake of bread for 3 weeks
Physical activity measured by the International Physical Activity Questionnaire (IPAQ) | 3 days
  Survey of participants' physical activities before and during the intake of bread for 3 weeks. The IPAQ contains 7 self-report questions and the categorical score is divided into 3 levels: low (less than 600 metabolic equivalent-minutes/week), moderate (at least 600 metabolic equivalent-minutes/week) or high (at least 1500 metabolic equivalent-minutes/week).
Quality of life measured by the Euro Quality of Life questionnaire | once before and after intake of bread for 3 weeks
  Survey of participants' well-being before and during the intake of bread for 3 weeks. It records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled from 0 (worst imaginable health state) to 100 (best imaginable health state).
Perceived stress measured by a Visual analog scale questionnaire | before the stress test, after the introduction phase, directly after the acute stress phase, 5 minutes, 10-15 minutes, 60 minutes, and 75 minutes after the stress test
  Difference in the perceived stress during a stress test between and within intervention groups after the intake of bread for 3 weeks
Cognitive control using Eriksen flanker task (Flanker task) | once before and after intake of bread for 3 weeks
  Difference in cognitive control between and within intervention groups after the intake of bread for 3 weeks
Working memory performance using a modified N-back task combined with recent-probes item-recognition task (Sternberg task) | once before and after intake of bread for 3 weeks
  Difference in working memory between and within intervention groups after the intake of bread for 3 weeks
Electrocardiogram (ECG) using the Biopac system | once before and after intake of bread for 3 weeks
  Difference in heart rate variability during a stress test between and within intervention groups after the intake of bread for 3 weeks
Electrodermal activity (EDA) using the Biopac system | once before and after intake of bread for 3 weeks
  Difference in skin conductivity during a stress test between and within intervention groups after the intake of bread for 3 weeks. Electrodes to measure EDA will be placed on the subjects' left palm. Skin conductivity measures will include skin conductivity level (SCL), the number of skin conductivity responses (SCR), and the amplitude of SCR.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Wall, PhD, Principal Investigator — Örebro University, Sweden
Locations (1):
- Örebro University, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: No